CLINICAL TRIAL: NCT01087047
Title: Upper Airways in Pregnancy: Evaluation by the Acoustic Reflection Method
Acronym: MAVAG
Status: Completed | Type: Observational
Sponsor: Club d'Anesthésie-Réanimation Pédiatrique Armand Trousseau (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Dr Nicolas LEBOULANGER, Dr, Club d'Anesthésie-Réanimation Pédiatrique Armand Trousseau
Other Study IDs: MAVAG
Record Dates: First submitted 2010-03-10; First posted 2010-03-15 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Pregnancy
Keywords: Pregnancy; Upper airways; Acoustic reflection method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Physiological modifications: Pregnant women who attend the routine ultrasound control in our institution before 14 weeks of pregnancy
  Interventions: Device: Acoustic reflection method
- MRI and acoustic: Women undergoing an MRI for obstetrical purpose
  Interventions: Device: Acoustic reflection method

INTERVENTIONS:
Device: Acoustic reflection method — An acoustic reflection device gives the longitudinal cross-sectional area profile along airways. It is based on the analysis of a planar acoustic wave propagating in a rigid duct connected to airway.

SUMMARY:
It is well known that airway management can be difficult during pregnancy. Increased risks for difficult intubation in pregnant women have been often reported. Thus, pregnancy is regarded as a period of high anesthesiologic risk.

Generalized weight gain is a well known factor influencing the upper airway in pregnant women. However, the modifications of the airway itself are less well documented.

The acoustic reflection method is based on the analysis of the reflection of a single transient planar wave allowing the analysis of the longitudinal cross-sectional area profile of the examined cavity. It is a noninvasive and harmless method.

The aim of the study is to evaluate by acoustic reflection method the physiological modifications of the upper airways during pregnancy.

Women enrolled in the study will undergo an acoustic recording during the first, second, and third trimester of pregnancy, as well as two days and one month after delivery. Forty pregnant women will be included in this monocentric, prospective, open labelled study.

Moreover, a single acoustic recording will be performed in 10 other pregnant women undergoing an MRI for obstetrical purpose. The estimated caliber of the upper airways by MRI and acoustic method will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who attend the routine ultrasound control in our institution before 14 weeks of pregnancy will be invited to participate in the study.
* Women are eligible for the study if they are:

  * healthy (no previous disease, hypertension, nor obesity),
  * 18 years or more
  * with a singleton live fetus at the routine ultrasound scan
  * with a normal pregnancy.

Exclusion Criteria:

* Pregnancy complications
* Multiple pregnancy
* High risk for preterm labor
* Underlying diseases that could interfere with the results (such as pre-existing upper airway problems) and participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Physiological modifications during pregnancy and acoustic reflection method | 6 months
  Main aim: to evaluate by acoustic reflection method the physiological modifications of the upper airways during pregnancy. Women enrolled in the study will undergo an acoustic recording during:
  * the 1st, 2d, and 3d trimester of pregnancy
  * two days after delivery
  * one month after delivery

SECONDARY OUTCOMES:
MRI and acoustic reflection method | 6 months
  Secondary aim: a single acoustic recording will be proposed to 10 pregnant women undergoing an MRI for obstetrical purpose.
  The estimated caliber of the upper airways by MRI and acoustic method will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte FAUROUX, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Nicolas LEBOULANGER, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Armand Trousseau University Hospital, Paris
  - Hôpital d'Enfants Armand Trousseau, Paris

REFERENCES:
- [Background] Kodali BS, Chandrasekhar S, Bulich LN, Topulos GP, Datta S. Airway changes during labor and delivery. Anesthesiology. 2008 Mar;108(3):357-62. doi: 10.1097/ALN.0b013e31816452d3. PMID 18292672
- [Background] Louis B, Fodil R, Jaber S, Pigeot J, Jarreau PH, Lofaso F, Isabey D. Dual assessment of airway area profile and respiratory input impedance from a single transient wave. J Appl Physiol (1985). 2001 Feb;90(2):630-7. doi: 10.1152/jappl.2001.90.2.630. PMID 11160063